CLINICAL TRIAL: NCT05747300
Title: Clinical and Radiographic Evaluation of Premixed Bioceramic Paste (Wellroot PT) Versus Mineral Trioxide Aggregate (MTA) in Pulpotomy of Primary Molars: A Randomized Clinical Pilot Study
Brief Title: Wellroot PT Versus MTA in Pulpotomy of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Gamal, Doaa Gamal Mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Experimental
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pulpotomy
Keywords: Pulpotomy wellroot PT bioceramic paste

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA pulpotomy (Active Comparator): Vital pulpotomy primary Molars using MTA
  Interventions: Other: Premixed bioceramic paste wellroot PT
- Wellroot PT pulpotomy (Experimental): Vital pulpotomy primary Molars using premixed bioceramic paste wellroot PT
  Interventions: Other: Premixed bioceramic paste wellroot PT

INTERVENTIONS:
Other: Premixed bioceramic paste wellroot PT — Vital pulpotomy primary Molars using premixed bioceramic paste wellrootPT
  Other Names: Wellroot PT

SUMMARY:
compare the clinical and radiographic success of mineral trioxide aggregate (MTA) versus premixed bioceramic paste (Wellroot PT) as pulpotomy medicaments in primary molars.

DETAILED DESCRIPTION:
Preservation of primary dentition decreases the risk of developing any occlusal abnormalities caused by premature loss of primary teeth, which are considered natural space maintainers for the successor permanent teeth, therefore vital pulp therapy is of a big concern in the research field in pediatric dentistry .

One of the most commonly used regenerative materials in pulpotomies is Mineral Trioxide Aggregate (MTA) which showed a high success rate clinically and radiographically when compared to other materials due to its biocompatibility, antibacterial properties and excellent sealing ability . However it has some drawbacks such as difficult manipulation and handling because it is supplied in powder and liquid form which need mixing. Mixing is operator dependant and may be not uniform if handled wrongly, technique sensitive, potential discoloration, and long setting time.

Premixed bioceramics Well-Root™ PT (Vericom, Gangwon-Do, Korea) have been introduced into the market and present with desirable properties as a pulp capping agent. Owing to good handling characteristics, biocompatibility, odontogenic property and antibacterial action, the premixed bioceramic materials are recommended for procedures such as pulp capping, pulpotomy, perforation repair, root-end filling, and obturation.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged between 4 years and 7 years.

  * Mandibular second primary molar with deep caries involving pulp.
  * No history of spontaneous pain, pathologic mobility, draining sinus tract, redness or swelling of the vestibule.
  * Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.

Radiographic criteria:

* No sign of radiolucency in periapical or furcation area.
* No widening of PDL space or loss of lamina dura continuity.
* No evidence of internal/external pathologic root resorption.

Exclusion Criteria:

* • Uncooperative children.

  * Children with systemic disease.
  * Lack of informed consent by the child patient's parent.
  * Unable to attend follow-up visits.
  * Refusal of participation.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 1 year
  Binary (present/absent) Verbal question to patient/ parent
Soft tissue pathology | 1 year
  Binary (present/absent) Visual clinical examination
Pain to percussion | 1 year
  Binary (present/absent) Percussion test by the back of the dental mirror
Pathologic mobility | 1 year
  Binary (present/absent) Mobility test (pressure using the end of two dental mirrors)

SECONDARY OUTCOMES:
Absence of furcation or periapical radiolucency Absence of external or internal root resorption | 1 year
  Binary (present/absent) Intraoral digital periapical X-ray